CLINICAL TRIAL: NCT03086928
Title: One Year Clinical Evaluation of E-max CAD and Lava Ultimate Laminate Veneers With Butt Joint Preparation
Brief Title: One Year Clinical Evaluation of E-max CAD and Lava Ultimate Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Eltohami, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-3-12
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Discoloration, Tooth
MeSH Terms: conditions — Tooth Discoloration | interventions — IPS e.max CAD LT

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lava ultimate (Experimental): lava ultimate is Resin nano-ceramic which is a mixture of a resin composite matrix and nano-ceramic fillers of approximately 80% by weight. The main advantages of this material over the glass ceramics are the stress absorbing action or stress distribution by having modulus of elasticity near to the tooth dentin and can be individualized intra-orally or extra-orally, either before or after definitive cementation.
  Interventions: Other: lava ultimate
- E.max cad (Active Comparator): E.max is lithium disilicate glass ceramic, composed of quartz, lithium dioxide, phosphor oxide, alumina oxide, and potassium oxide with superior mechanical and optical properties if used for laminate veneers
  Interventions: Other: E.max cad

INTERVENTIONS:
Other: lava ultimate — resin nano ceramic material
  Arms: lava ultimate
Other: E.max cad — Lithium disilicate glass ceramic
  Arms: E.max cad

SUMMARY:
Restoration of anterior teeth using conservative approach allows clinicians to provide porcelain laminate veneers with excellent esthetics without extensive tooth structure removal. laminate veneers need the use of etch-able ceramics like glass ceramics (E.max) and hybrid ceramics (Lava Ultimate). The aim of this study is to compare both e.max and lava ultimate veneers clinically.

DETAILED DESCRIPTION:
The use of E-max CAD well documented in the literatures as successful restoration modality which has superior optical and mechanical properties. The introduction of hybrid ceramic materials combined the advantages of both glass ceramics and composite resin. Resin nano-ceramic is a mixture of a resin composite matrix and nano-ceramic fillers of approximately 80% by weight. The main advantages of this material over the glass ceramics are the stress absorbing action or stress distribution by having modulus of elasticity near to the tooth dentin and can be individualized intra-orally or extra-orally, either before or after definitive cementation.

Yet there are no studies for clinical evaluation of both mentioned laminate veneers restorations. This study is conducted to compare between both materials clinically according to modified USPHS criteria in terms of marginal adaptation, fracture, debonding, marginal discoloration and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Be physically and psychologically able to tolerate conventional restorative procedures.
3. Have no active periodontal or pulpal diseases, have teeth with good restorations.
4. Patients with teeth problems indicated for laminate veneer (e.g. discoloration, defect not involve more than 60% enamel loss, mild malposition, anterior upper….).
5. Be willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patient with fractured teeth of more than 60% enamel loss.
3. Patients with poor oral hygiene and motivation.
4. Pregnant women.
5. Psychiatric problems or unrealistic expectations.
6. Lack of opposite occluding dentition in the area intended for restoration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction evaluated by using a questionnaire | one year
  Patient satisfaction will be evaluated by using a questionnaire, which will be translated. A validation of the Arabic translation will be done before using the questionnaire in the trial. Each participant will take the questionnaire into a quiet room and will be left alone until questionnaire is totally answered.

SECONDARY OUTCOMES:
Modified USPHS criteria | one year
  It is a criteria for clinical evaluation of dental restorative materials in terms of marginal adaptation, marginal discoloration, fracture, debonding.

CONTACTS AND LOCATIONS:
Overall Officials: amina zaki, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pimentel W, Teixeira ML, Costa PP, Jorge MZ, Tiossi R. Predictable Outcomes with Porcelain Laminate Veneers: A Clinical Report. J Prosthodont. 2016 Jun;25(4):335-40. doi: 10.1111/jopr.12413. Epub 2015 Dec 3. PMID 26633080
- [Background] D'Arcangelo C, De Angelis F, Vadini M, D'Amario M. Clinical evaluation on porcelain laminate veneers bonded with light-cured composite: results up to 7 years. Clin Oral Investig. 2012 Aug;16(4):1071-9. doi: 10.1007/s00784-011-0593-0. Epub 2011 Jul 20. PMID 21773711